CLINICAL TRIAL: NCT02426684
Title: A Phase I/II Trial to Evaluate the Safety and Tolerability of Ides® (IgG Endopeptidase) to Eliminate Donor Specific HLA Antibodies (DSAs) and Prevent Antibody-Mediated Rejection Post-Transplant in Highly-HLA Sensitized Patients.
Brief Title: Ides in Highly Sensitized (HS) Patients Awaiting Kidney Transplantation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: Hansa Biopharma AB (Industry)
Responsible Party: Principal Investigator, Stanley Jordan, MD, MD, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IdeSCSMC
Record Dates: First submitted 2015-04-22; First posted 2015-04-27 (Estimated); Results first posted 2022-05-16 (Actual); Last update posted 2022-05-16 (Actual); Status verified 2022-04

CONDITIONS: Renal Disease
Keywords: End Stage Renal Disease; Kidney Transplant; Desensitization; Highly Sensitized; Antibodies
MeSH Terms: conditions — Kidney Diseases; Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IdeS® (Experimental): Twenty patients will receive 0.24mg/kg (n=20)
  Interventions: Drug: IdeS® (Imlifidase)

INTERVENTIONS:
Drug: IdeS® (Imlifidase) — 0.24mg/kg IdeS
  Other Names: IgG endopeptidase

SUMMARY:
This is a single center phase I/II open label, exploratory study assessing safety and efficacy of IdeS® (Hansa Medical, Lund, Sweden) given immediately prior to kidney transplantation. We hope that IdeS® will help eliminate DSAs in HS patients who are DSA+ and flow cytometry (FCMX) crossmatch + at time of transplant. We plan to enroll a total of 20 patients. Patients will be followed for 6 months post administration of IdeS®.

DETAILED DESCRIPTION:
IdeS® is an IgG-degrading enzyme of S.pyogenes that cleaves all four human subclasses of IgG with strict specificity. Alloantibodies are a major deterrent to access to and success of life-saving organ transplants. We hypothesize that the use of IdeS® pre-transplant in HS patients will represent a more robust and complete technique to eliminate DSA from the sera of HS patients. A single dose administration of IdeS® in the pre-operative period to HS patients with positive DSAs and flow cytometry crossmatches will durably eliminate circulating DSAs, allow transplantation to occur without ABMR and, in conjunction with standard desensitization therapy, result in a durable suppression of DSA levels thus eliminating the risk for ABMR.

ELIGIBILITY:
Inclusion Criteria:

* End-stage renal disease awaiting transplantation on the UNOS list.
* No known contraindications for therapy with IVIG10%/Rituximab, plasmapheresis (PLEX) or IdeS®.
* Age 18-70 years at the time of screening.
* Calculated PRA (CPRA)> 50% demonstrated on 3 consecutive samples, Patient highly-HLA sensitized and a candidate for DD transplantation after desensitization at CSMC.
* At transplant, patient must have donor-specific antibody/ crossmatch positive (DSA/CMX+) non-HLA identical donor.
* Pre-transplant vaccination with Streptococcus pneumoniae and Nisseria meningitides
* Subject/Parent/Guardian must be able to understand and provide informed consent.

Exclusion Criteria:

* Positivity for anti-IdeS IgE
* Use of IVIG 4 weeks prior to planned IdeS® administration
* Recipients of Extended Criteria Donors (ECD) or Living Donors (LD)
* Lactating or pregnant females.
* Women of child-bearing age who are not willing or able to practice FDA-approved forms of contraception.
* HIV-positive subjects.
* Subjects who test positive for HBV infection [positive HBVsAg, HBVcAb, or HBVeAg/DNA] or HCV infection [positive Anti-HCV (EIA) and confirmatory HCV RIBA].
* Subjects with active TB.
* Subjects with selective IgA deficiency, those who have known anti-IgA antibodies, and those with a history of anaphylaxis or severe systemic responses to any part of the clinical trial material.
* Subjects who have received or for whom multiple organ transplants are planned.
* Recent recipients of any licensed or investigational live attenuated vaccine(s) within two months of the screening visit (including but not limited to any of the following:

  1. Adenovirus [Adenovirus vaccine live oral type 7]
  2. Varicella [Varivax]
  3. Hepatitis A [VAQTA]
  4. Rotavirus [Rotashield]
  5. Yellow fever [Y-F-Vax]
  6. Measles and mumps [Measles and mumps virus vaccine live]
  7. Measles, mumps, and rubella vaccine [M-M-R-II]
  8. Sabin oral polio vaccine
  9. Rabies vaccines [IMOVAX Rabies I.D., RabAvert])
* A significantly abnormal general serum screening lab result defined as a WBC < 3.0 X 103/ml, a Hgb < 8.0 g/dL, a platelet count < 100 X 103/ml, , an SGOT > 3X upper limit .
* Individuals deemed unable to comply with the protocol.
* Subjects with active CMV or EBV infection as defined by CMV-specific serology (IgG or IgM) and confirmed by quantitative PCR with or without a compatible illness.
* Subjects with a known history of previous myocardial infarction within one year of screening.
* Subjects with a history of clinically significant thrombotic episodes, and subjects with active peripheral vascular disease.
* Subjects with Protein C and Protein S deficiency
* Use of investigational agents within 4 weeks of participation.
* Known allergy/sensitivity to IdeS® infusions

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2015-06-16 (Actual); Primary Completion 2017-11-10 (Actual); Study Completion 2017-11-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stanley C Jordan, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

REFERENCES:
- [Background] von Pawel-Rammingen U. Streptococcal IdeS and its impact on immune response and inflammation. J Innate Immun. 2012;4(2):132-40. doi: 10.1159/000332940. Epub 2012 Jan 17. PMID 22248585
- [Derived] Jordan SC, Lorant T, Choi J, Kjellman C, Winstedt L, Bengtsson M, Zhang X, Eich T, Toyoda M, Eriksson BM, Ge S, Peng A, Jarnum S, Wood KJ, Lundgren T, Wennberg L, Backman L, Larsson E, Villicana R, Kahwaji J, Louie S, Kang A, Haas M, Nast C, Vo A, Tufveson G. IgG Endopeptidase in Highly Sensitized Patients Undergoing Transplantation. N Engl J Med. 2017 Aug 3;377(5):442-453. doi: 10.1056/NEJMoa1612567. PMID 28767349

RESULTS

PARTICIPANT FLOW:
Groups:
- IdeS® 0.24mg/kg: Twenty patients were planned to receive 0.24mg/kg (n=20). 17 patients in total were enrolled in this study. The study closed to enrollment before completing the intended 20 participant enrollment; with 3 allocations remaining.
Period: Overall Study
Arm/Group | IdeS® 0.24mg/kg
Started | 17
Completed | 16
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Groups:
- IdeS® 0.24 mg/kg: patients who received 0.24mg/kg (n=17)
Arm/Group | IdeS® 0.24 mg/kg
Number analyzed (Participants) | 17
Age, Customized [Mean (Standard Deviation); unit: years] | 41.6 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Allograft Rejection
Description: Number of participants with allograft rejection will be assessed at 6 month post transplant renal biopsy.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | IdeS® 0.24 mg/kg
Number analyzed (Participants) | 13
Participants | 7

2. Secondary Outcome: eGFR
Description: eGFR based on serum creatinine will be collected 6 months post transplant.
Time Frame: 6 months post transplant
Measure: Mean (Standard Deviation); unit: ml/min/m2
Arm/Group | IdeS® 0.24 mg/kg
Number analyzed (Participants) | 13
ml/min/m2 | 66 (48)

3. Secondary Outcome: Proteinuria
Description: Urine total protein & urine creatinine will be drawn from day 0 to day 30, and urinalysis will be collected on day 180 from transplant.
Time Frame: 6 months post transplant
Population: This outcome was not assessed
Arm/Group | IdeS® 0.24 mg/kg
Number analyzed (Participants) | 0

4. Secondary Outcome: Number of Participants With Donor Specific Antibodies (DSA) Post-transplant
Description: Donor specific antibody levels will be checked at Day 180 post transplant to see if patients developed new antibodies or antibody intensity levels worsened post transplant. The DSA mean fluorescence intensity (MFI) was recorded, in comparison to the levels at transplant. This outcome measure was intended to record if any of the participants had a new DSA formation at Day 180, or if any participant had higher MFI levels of the DSA at Day 180, compared to baseline.
Time Frame: 6 months post transplant
Measure: Count of Participants; unit: Participants
Arm/Group | IdeS® 0.24 mg/kg
Number analyzed (Participants) | 14
Participants | 4

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | IdeS® 0.24 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/17
Serious Adverse Events (participants affected / at risk) | 5/17
Other Adverse Events (participants affected / at risk) | 0/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IdeS® 0.24 mg/kg (N=17)
Infection (UTI) (Infections and infestations) | 2 (2)
Malignant hyperthermia (General disorders) | 1 (1)
Fever and anemia (Blood and lymphatic system disorders) | 1 (1)
moderate hydronephrosis and ureteral obstruction (Renal and urinary disorders) | 1 (1)
abdominal pain, nausea, vomitting (Gastrointestinal disorders) | 2 (2)
Elevated Cr and Afib with RVR after peritneal dialysis (Renal and urinary disorders) | 1 (1)
CHF exacerbation and AKI (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-24): https://cdn.clinicaltrials.gov/large-docs/84/NCT02426684/Prot_SAP_001.pdf